CLINICAL TRIAL: NCT03916692
Title: Glycemic Response of Amylopectin Containing Drinks
Brief Title: GRAPE • Glycemic Response of Amylopectin Containing Drinks
Acronym: GRAPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 restrictions
Sponsor: Arizona State University (Other)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00016578
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Glycemic Index

STUDY DESIGN:
Intervention Model Description: Randomized Cross-over trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Process - glucose balance (Experimental): Standard Process - glucose balance formula (200 kcal)
  Interventions: Dietary Supplement: Carbohydrate drink
- Energy smart Carbohydrate blend (Experimental): Energy smart carbohydrate blend (50 grams, 200 kcal)
  Interventions: Dietary Supplement: Energy smart Carbohydrate blend
- Liquid Dextrose Control (Active Comparator): Liquid dextrose solution in the form of TRUTOL ® Glucose Tolerance Test Beverage (50 grams, 200 kcal)
  Interventions: Dietary Supplement: Liquid Dextrose

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink — Meal replacement drink containing 200 kcal
  Other Names: SP-glucose balance formula
  Arms: Standard Process - glucose balance
Dietary Supplement: Energy smart Carbohydrate blend — Carbohydrate blend drink designed for low glycemic responses containing 200 kcal
  Arms: Energy smart Carbohydrate blend
Dietary Supplement: Liquid Dextrose — Liquid Dextrose drink of 200 kcal
  Arms: Liquid Dextrose Control

SUMMARY:
To quantify the glycemic index of the SP energy-smart-based nutrition supplement and the SP Glucose-support formula as compared to a glucose drink. We hypothesized that both the energy-smart-based nutritional supplement and the SP Glucose-support formula will have low glycemic index.

The aim of the study is to quantify the glycemic index of the SP energy-smart-based nutrition supplement and the SP Glucose-support formula as compared to a glucose drink. We hypothesized that both the energy-smart-based nutritional supplement and the SP Glucose-support formula will have low glycemic index.

DETAILED DESCRIPTION:
Subjects: 9 non-diabetic (HbA1c < 6.5) males aged 30-55 years with body mass indices ranging from 27.5 to 35 kg∙m-2. Individuals with impaired glucose tolerance will be included as long as they are not diagnosed with diabetes and their HbA1c is less than 6.5.

Preliminary Testing: Medical history, weight, height, body composition via dual x-ray absorptiometry (DXA) and glycosylated hemoglobin (HbA1c) measurement.

Protocol: After a 10-hour overnight fast, subjects will complete 3 experimental visits in which they will ingest one of three beverages in a randomized order. During experimental visits subjects will either be given the following 3 experimental drinks:

* Full SP-glucose balance formula (200 kcal)
* Energy smart carbohydrate blend (50 g, 200 kcal)
* Liquid dextrose solution in the form of TRUTOL ® Glucose Tolerance Test Beverage (50 g, 200 kcal)

ELIGIBILITY:
Inclusion Criteria:

* BMI 27.5 to 35 kg∙m-2

Exclusion Criteria:

* Diagnosed diabetes
* HbA1c > 6.5
* competitive athletes
* body weigh change > 3kg during last month

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-reported
Enrollment: 15 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve of Glucose | 120 minutes
  Positive integer of the area under the Curve of glucose
Area Under the Curve for Insulin | 120 minutes
  Positive integer of the area under the Curve of insulin
Blood glucose | 30, 60 and 120 minutes of the glucose challenge
  Blood glucose levels
Blood insulin | 30, 60 and 120 minutes of the glucose challenge
  Blood insulin levels

SECONDARY OUTCOMES:
c-peptide | 30, 60, and 120 minutes of the glucose challenge
  Blood levels of c-peptide
glucagon | 30, 60, and 120 minutes of of the glucose challenge
  Blood levels of glucagon
Leptin | 30, 60, and 120 minutes of the glucose challenge
  Blood levels of leptin
Adiponectin | 30, 60, and 120 minutes of the glucose challenge
  Blood levels of adiponectin
glucagon-like-peptide-1 | 30, 60, and 120 minutes of the glucose challenge
  Blood levels of glucagon-like-peptide-1

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Kavouras, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No